CLINICAL TRIAL: NCT04759742
Title: The Optimal Dosage of Ropivacaine for Arthroscopic Knee Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yanchao Yang (Other)
Responsible Party: Sponsor-Investigator, Yanchao Yang, Principal investigator, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Arthroscopic anesthesia
Record Dates: First submitted 2021-02-07; First posted 2021-02-18 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Arthroscopic Knee Surgery; Ropivacaine; Combined Spinal Epidurai Anesthesia; ED50; ED95
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group Ropivacaine (Experimental): The recommended administration concentration of ropivacaine in the subarachnoid space was 0.5% and the dose was 2-3ml (practical clinical anesthesiology). Based on previous clinical experience, the starting dose of ropivacaine was set at 12.5mg (2.5ml) and Dixon's up-and down method was adopted (Dixon WJ, Massey FJ Jr. Introduction to Statistical Analysis. NY: McGraw-Hill;1969. P. 344.) The dose of ropivacaine in the next patient was adjusted to 0.5mg (0.1 mL) according to the results of the previous patient's trial.
  Interventions: Drug: ropivacaine

INTERVENTIONS:
Drug: ropivacaine — According to previous clinical experience, 0.5% ropivacaine was given in the subarachnoid cavity, and the initial dose was set at 2.5 mL (12.5mg). Dixon's up-and down method was adopted to adjust or down-adjust the dose of ropivacaine in the next patient according to the experimental results of the previous patient, and the adjusted dose was 0.1 mL (0.5mg).

SUMMARY:
Fast-track Surgery (FTS ) refers to the application of various proven effective methods in perioperative period to reduce stress and complications and accelerate the recovery of patients.Nowadays, FTS has been successfully applied in clinical practice."FTS" truly embodies the concept of "patient-centered" and the direction of medical development.

Lower limb joint damage (the meniscus, and patellar ligament, etc.) is the joint movement orthopedic common disease, often characterized by joint swelling, pain, sports relaxation instability, thigh muscle atrophy, most can't continue to pursue the original movement, even unbend and flexor limited activity, result in patients with walking difficulties, serious impact on the patient's quality of life.Practice has proved that minimally invasive surgery under arthroscopy is the best way to treat such injuries. According to literature reports, the average hospital stay after arthroscopy is 5~7 days, while successful application of FTS can shorten it to 2~3 days.

Anesthesia plays an important role in the process of FTS.Compared with general anesthesia, intra-spinal anesthesia can effectively reduce the incidence of postoperative complications in patients, such as ventilator-related lung injury, deep vein thrombosis, cardiovascular and cerebrovascular accidents, and acute renal failure.Ropivacaine is a long-acting amide local anesthetic. Compared with bupivacaine, it is more and more widely used in spinal anesthesia due to its advantages of lower degree of motor nerve block and weaker toxicity to central nervous system and cardiac.However, the optimal dosage of ropivacaine for arthroscopic surgery is still unclear. Conventional dosage makes patients unable to move 2-4h after surgery and unable to urinate autonomically. Therefore, this study aims to optimize the dosage of ropivacaine for spinal anesthesia and enable patients to recover motor function at an early stage.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective arthroscopic knee surgery

  * ASA: grade I to III

Exclusion Criteria:

* There are contraindications to spinal anesthesia

  * Allergic to local anesthetics

    * Patient refused

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
the median effective dose (ED) of ropivacaine in knee arthroscopic surgery | from preoperative to postoperative 24 hours
  The primary outcome of this present study was the median effective dose (ED) of ropivacaine in knee arthroscopic surgery to allow immediate postoperative mobilization as well as adequate anesthesia during surgery.The up and down method as described by Dixon and Massey was used.This is a sequential allocation model in which patients received a dose of ropivacaine according to the outcome of the preceding patient. A starting dose of the test sequence was set to 12.5 mg ropivacaine .The dose of ropivacaine in the next patient was increased or decreased according to the experimental results of the previous patient, and the adjusted dose was 0.5mg.

CONTACTS AND LOCATIONS:
Overall Officials: junchao Zhu, Study Chair — Shengjing Hospital
Locations (1):
- Shengjing Hospital, Shengyang, Liaoning, China